CLINICAL TRIAL: NCT07117656
Title: Developing and Pilot Testing Project Vuselela for ART and OST Engagement in Johannesburg, South Africa
Brief Title: Project Vuselela Feasibility
Acronym: PV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11194429; R34DA062367 (NIH)
Record Dates: First submitted 2025-07-15; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: HIV; Drug Users
MeSH Terms: conditions — Drug Misuse

STUDY DESIGN:
Intervention Model Description: Pilot study to understand intervention feasibility and preliminary impact on HIV and OST outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Four sessions on coping and communication skills to improve support for treatment among family members and people who inject drugs.
  Interventions: Behavioral: Project Vuselela
- Standard of Care (No Intervention): Offered current harm reduction services at clinics.

INTERVENTIONS:
Behavioral: Project Vuselela — A four session intervention with people who inject drugs and family members. Delivered three group sessions and one dyad session. Session content designed to improve coping and communication skills that will in turn improve treatment outcomes.
  Arms: Intervention

SUMMARY:
To develop an intervention that engages family members in supporting HIV and opioid substitution therapy treatment for those who inject drugs in South Africa, and then conduct a pilot study to understand feasibility and preliminary impact on outcomes.

DETAILED DESCRIPTION:
In response to increased injection drug use in Johannesburg, South Africa, and low ART and OST treatment retention rates, we will develop and pilot-test the intervention, Project Vuselela. The intervention is designed to engage family members in treatment support using a multi-session skill-building approach that is led by trained peer navigators. Both PLWHIDs and their family members will attend sessions to develop these skills and treatment action plans, facilitated by peer navigators. We will assess PLWHID and family acceptability of the intervention and preliminary impact on PLWHID ART and OST treatment adherence when compared to those in the current program as standard of care. The study will be conducted at Yeoville Clinic in Johannesburg, a setting with high rates of injection drug use and the only OST clinic in the city.

ELIGIBILITY:
Inclusion Criteria:

Aim 2 PLHWID Inclusion Criteria

1. Any sex or gender
2. >18 years of age
3. HIV-positive as per medical record
4. Self-reported injection drug use behavior
5. Have not participated in the current ART-OST program
6. Initiating ART or OST
7. Identifies a potential family member who can provide support
8. Live in Johannesburg

Family Member Inclusion Criteria

1. 18 years of age or older
2. Confirms family member (parent, sibling, partner, aunt, uncle, grandparent, cousin)
3. Knowledge of the drug using behavior by the PLWHID, but knowledge of their HIV status is not required.
4. No recent history of self-reported drug-using behavior (< 5 years)

Exclusion Criteria:

PLHWID Exclusion Criteria

1. Under 18 years of age
2. HIV-negative as per medical record
3. Notself-reported injection drug use behavior
4. Has participated in the current ART-OST program
5. Taking ART or OST
6. Cannot identify a potential family member who can provide support
7. Does not live in Johannesburg

Family Member Exclusion Criteria

1. Under 18 years of age
2. Not a family member
3. Does not know about drug using behavior by the PLWHID
4. Recent history of self-reported drug-using behavior (< 5 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2027-08-28 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | 3 and 6 months
  Assess feasibility, acceptability, willingness and safety. This will be completed using in-depth interviews and a study-specific survey.
Antiretroviral Therapy Therapy (ART) Adherence | 3 and 6 months
  Medical chart review of monthly anti-retroviral therapy (ART) prescription refill data will be collected. ART is medication to manage HIV infection.
Opioid Substitution Therapy (OST) Adherence | 3 and 6 months
  Medical chart review of opioid substitution therapy (OST) pick-up. This measure assesses use of OST to reduce effects of addiction.

CONTACTS AND LOCATIONS:
Locations (1):
- Anova Health Institute, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided